CLINICAL TRIAL: NCT00425191
Title: A Multicenter, Randomized Phase II Study Evaluating the Feasibility and Activity of Two Different Combinations of Docetaxel and Gemcitabine and of Cisplatin/Gemcitabine Followed by Docetaxel as First Line Therapy for Locally Advanced Unresectable or Metastatic Non-small Cell Lung Cancer.
Brief Title: Taxotere Combinations as First Line Therapy for Locally Advanced Unresectable or Metastatic Non-small Cell Lung Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XRP6976B_2501
Record Dates: First submitted 2007-01-19; First posted 2007-01-22 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Gemcitabine

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Docetaxel and Gemcitabine
- 2 (Experimental)
  Interventions: Drug: Docetaxel and Gemcitabine
- 3 (Experimental)
  Interventions: Drug: Gemcitabine cisplatin followed by docetaxel

INTERVENTIONS:
Drug: Docetaxel and Gemcitabine — Docetaxel: 40 mg/m², administered IV over 60 minutes (infusion drop by drop during the first five minutes) on day 1 and 8 immediately followed by Gemcitabine: 1200 mg/m2, administered IV over 30 minutes on day 1 and 8
  Arms: 1
Drug: Docetaxel and Gemcitabine — Docetaxel: 50 mg/m², administered IV over 60 minutes (infusion drop by drop during the first five minutes) on day 1 and 15 immediately followed by Gemcitabine: 1600 mg/m2, administered IV over 30 minutes on day 1 and 15.
  Arms: 2
Drug: Gemcitabine cisplatin followed by docetaxel — Gemcitabine: 1200 mg/m2, administered IV over 30 minutes on day 1 and 8 followed by Cisplatin 75 mg/m2, administered IV over 30-60 minutes on day 2
  Arms: 3

SUMMARY:
To assess the antitumour activity (response rate) in patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) of two different combinations of docetaxel and gemcitabine and of a sequential treatment of cisplatin /gemcitabine followed by docetaxel as first line chemotherapy · To evaluate the quantitative and qualitative toxicity of each treatment arms.· To determine time to progression, duration of response, time to treatment failure, and overall survival in each group.· To evaluate changes from baseline in the Lung Cancer Symptom Scale of patients in each treatment arm.

ELIGIBILITY:
The following information on clinical trials is provided for information purposes only to allow patients and physicians to have an initial discussion about the trial. This information is not intended to be complete information about the trial, to contain all considerations that may be relevant to potential participation in the trial, or to replace the advice of a personal physician or health professional.

Main criteria are listed hereafter:

Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of NSCLC istologic subtypes may include large cell, squamous cell, or adenocarcinoma or a generic cytological diagnosis of NSCLC;
* Patients must have a locoregionally advanced unresectable non metastatic NSCLC Stage IIIB (only N3 supraclavicular or T4 for pleural effusion) or Stage IV according to the revised International Staging System
* Patients must have at least one measurable lesion;
* Previous radical surgery (more 30 days before study entry) is allowed but a pathologic proof of progression of neoplastic disease must be documented whenever possible;
* Weight loss < = 5% within the last 3 months;
* Laboratory requirements at entry :

  * Blood cell counts: Absolute neutrophils > 2.0 x 109/LPlatelets > 100 x 109/LHemoglobin > 10 g/dl
  * Renal function:Serum creatinine < 1 upper normal limits (UNL). In case of limit value of serum creatinine, the creatinine clearance should be > 60 mL/min
  * Hepatic functions:Serum bilirubin < 1 x UNLASAT and ALAT < 2.5 x UNLAlkaline phosphatase < 5 x UNL (unless accompanied by extensive bone metastases);

Exclusion criteria:

* Prior systemic chemotherapy or immunotherapy including neoadjuvant or adjuvant treatments;
* Prior radiotherapy for NSCLC;
* Cyto-histological diagnosis of small cell lung cancer, carcinoid, or mixed small-cell / non-small cell lung cancer;
* Patients with not measurable disease only;
* Patients with symptomatic brain metastases or with leptomeningeal disease. However; patients with symptomatic brain metastases who become asymptomatic under corticosteriods treatment can enter the study;
* History of prior malignancies, except for cured non melanoma skin cancer, curatively treated in situ carcinoma of the cervix or other cancer curatively treated and with no evidence of disease for at least five years;
* History of hypersensitivity reaction to polysorbate 80;
* Pregnant or lactating women (women of childbearing potential must use adequate contraception);
* Concurrent treatment with other experimental drugs;
* Current peripheral neuropathy NCI grade > = 2;
* Significant neurological or psychiatric disorders;
* Hepatic functions abnormalities;
* Participation in clinical trials with other experimental agents within 30 days of study entry;
* Other serious concomitant illness of medical conditions;
* History of significant neurologic or psychiatric disorders including demential or seizures;
* Active infection requiring iv antibiotics;
* Active ulcer, unstable diabetes mellitus or other contra-indication to corticotherapy;
* Any other condition, which in the judgement of the investigator would place the subject at, undoes risk or interferes with the study.
* Treatment with biphosphonates.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2002-07; Primary Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Response Rate | Performed after 3 cycles and at the end of treatment (6 cycles).

SECONDARY OUTCOMES:
Time to progression. | Time from treatment to the documented profession of disease.

CONTACTS AND LOCATIONS:
Overall Officials: Georges Paizis, MD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Milan, Italy